CLINICAL TRIAL: NCT04835675
Title: Development and Validation of the Performance of a cfDNA Methylation-based Model Combined With Serum Tumor Markers for Early Hepatobiliary Malignancies Detection
Brief Title: AssesSment of Early-deteCtion basEd oN liquiD Biopsy in Hepatobiliary Cancer Malignancies
Acronym: ASCEND-Hep
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangzhou BR (Unknown)
Responsible Party: Sponsor
Other Study IDs: ZJYY-2020006
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2021-04

CONDITIONS: Hepatobiliary Malignancies
Keywords: Hepatobiliary malignancies; Liquid biopsy; Cell-free DNA; Early detection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Arm: Participants with new diagnosis of hepatobiliary malignancies, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test
- Benign Diseases Arm: Participants with benign diseases of the hepatobiliary system, from whom blood samples will be collected
  Interventions: Device: Multi-cancer early detection test

INTERVENTIONS:
Device: Multi-cancer early detection test — Blood collection and multi-cancer early detection testing

SUMMARY:
This study is a prospective, multicenter study aimed to develop and validate the performance of combined assays for cfDNA methylation markers and serum tumor markers in early hepatobiliary malignancies detection. Circulating tumor DNA (ctDNA) mutation, blood RNA markers and tissue will also be evaluated. The study will enroll approximately 496 participants, including participants with malignant or benign diseases of the hepatobiliary system.

ELIGIBILITY:
Inclusion Criteria for All the Participants:

* 40-75 years old
* Ability to comply with study procedures
* Ability to provide a written informed consent

Exclusion Criteria for All the Participants:

* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Recipients of anti-microbial therapy within 14 days prior to study blood draw
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer

Inclusion Criteria for Cancer Arm Participants:

* Confirmed diagnosis or highly suspicious cases of hepatobiliary malignancies
* No prior or ongoing anti-cancer therapy (local or systematic) prior to study blood draw

Exclusion Criteria for Cancer Arm Participants:

* Current diagnosis of other malignancies or multiple primary tumors
* Diagnosis of benign diseases by histopathological assessments
* Inability to characterize whether the lesion is malignant or benign
* Prior or ongoing treatment of cancer

Inclusion Criteria for Benign Diseases Arm Participants:

* Confirmed diagnosis of benign diseases of the hepatobiliary system
* No prior radical treatment of the benign diseases prior to study blood draw

Exclusion Criteria for Benign Diseases Arm Participants:

* Current or history of malignancies or precancerous lesions
* No confirmed diagnosis or inability to characterize a benign disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and assigned into two arms, including participants with new diagnosis of hepatobiliary malignancies and benign diseases of the hepatobiliary system.
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of early hepatobiliary malignancies detection and Tissue of origin (TOO) accuracy of a cfDNA methylation-based model combined with serum tumor markers when specificity was 90%, 95% or 98% | 16 months
Sensitivity and specificity of early hepatobiliary malignancies detection and TOO accuracy of a cfDNA methylation-based model combined with serum tumor markers | 16 months

SECONDARY OUTCOMES:
Sensitivity and specificity of a cfDNA methylation-based model combined with serum tumor markers in early detection of hepatobiliary malignancies in different stages | 16 months
Sensitivity and specificity of a cfDNA methylation-based model combined with serum tumor markers, clinical characteristics and other biomarkers | 16 months
Sensitivity and specificity of a cfDNA methylation-based model combined with serum tumor markers in participants with malignant or benign diseases of the hepatobiliary system | 16 months
Sensitivity and specificity of a cfDNA methylation-based model or serum tumor markers in participants with hepatobiliary malignancies | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Mingxin Pan, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No